CLINICAL TRIAL: NCT05264714
Title: Cluster Headache Treatment With Rimegepant-Open Label Pilot Study
Brief Title: Cluster Headache Treatment With Rimegepant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Carrie (Beth) E. Robertson, MD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-003394
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — rimegepant sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cluster Headache Subjects (Experimental): Subjects with cluster headaches will track their headaches for a one-week baseline headache diary. After establishing the baseline headache frequency, severity, and abortive medicine use, subjects will be asked to start their first dose of rimegepant with their next moderate to severe cluster headache.
  Interventions: Drug: Rimegepant

INTERVENTIONS:
Drug: Rimegepant — 150 mg oral disintegrating tablet every other day for one week
  Other Names: Nurtec ODT

SUMMARY:
The purpose of this research is to explore the efficacy of rimegepant as a preventative therapy for cluster headache.

DETAILED DESCRIPTION:
This is a prospective, open-label pilot study to investigate the use of rimegepant for the treatment of cluster headache. Subjects will be screened at outpatient clinic visit appointments and interested qualified subjects will be consented and offered participation in this trial. Once consent has been obtained, patients with cluster headache will start immediately keeping track of their headaches for a one-week baseline. In contrast, patients with episodic cluster headache will be asked to contact the study coordinator at the onset of their next cluster cycle, at which point they will repeat the screening and then start their one-week baseline headache diary. After establishing the baseline headache frequency, severity, and abortive medicine use, patients will be asked to start their first dose of study drug with their next moderate to severe cluster headache. They will rate their pain for this headache on a 5 point severity scale ("no headache," "mild," "moderate," "severe" or "very severe" and rate the pain on a scale of 0 to 10 ("0" is no pain and "10" is most severe pain imaginable) at the time of taking rimegepant and rate the pain again at 15, 30, 45, and 60 minutes after taking the drug. 60 or more minutes after taking the rimegepant, they are allowed to use their usual standard of care for the acute/abortive treatment of acute cluster attacks. After this first dose, they will then take rimegepant on an every other day schedule for a total of 4 doses over 8 days. A final visit for evaluation and collection of headache diaries will be conducted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of recurrent cluster headaches, as described by ICHD-3 (International Classification of Headache Disorders-3):

  * Severe or very severe unilateral orbital, supraorbital and/or temporal pain lasting 15-180 minutes, when untreated.
  * Headache is accompanied by at least one of the following:

    * Ipsilateral conjunctival injection and/or lacrimation;
    * Ipsilateral nasal congestion and/or rhinorrhea;
    * Ipsilateral eyelid edema;
    * Ipsilateral forehead and facial sweating;
    * Ipsilateral miosis and/or ptosis;
    * A sense of restlessness or agitation.
  * Headache attacks occur at a frequency between every other day and 8 per day.
  * Headaches are not attributed to another disorder.
* Subjects able to distinguish cluster headache attacks from other headache disorders, such as migraine.
* Subjects on prophylactic headache medicines other than verapamil will be permitted to remain on these with possible headache-prophylactic effects if the dose is stable for at least 2 months (onabotulinumtoxinA injections stable for 6 months) prior to the screening visit and the dose is not expected to change during the course of the study.
* Prior MR (magnetic resonance) imaging of head (CT if MRI contraindicated) performed after the onset of headaches.
* Subjects agree to refrain from starting a new prophylactic cluster headache medicine, including steroids and nerve blocks, during the course of the study.
* Subjects are required to have a cluster headache attack fre-quency ranging from one attack every other day to eight attacks per day, with at least four total attacks during the one-week prospective baseline period. Additionally, episodic cluster headache patients are required to have a history of cluster head-ache period lasting at least 6 weeks.

Exclusion Criteria:

* Subjects with a history of an adverse reaction to CGRP (calcitonin gene-related peptide) antibodies or another CGRP antagonist (gepant).
* Subjects with episodic cluster who are felt to be toward the end of their cluster cycle (estimated to be within the last 4 weeks).
* Pregnancy (negative serum pregnancy testing at enrollment and use of contraception considered to be effective).
* Subjects with a history of uncontrolled, unstable, or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Subjects with myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery bypass graft (CABG), stroke, or transient ischemic attack (TIA) in the 6 months prior to screening.
* Subjects with other pain syndromes, psychiatric conditions, dementia or significant neurological disorders that, in the investigator's opinion might interfere with study assessments.
* Use of peripheral nerve blocks (e.g., occipital, supraorbital, auriculotemporal, and/or sphenopalatine ganglion nerve blocks) one month prior to enrollment.
* Use of opioids or barbiturates more than 5 days per month.
* Use of other small molecule CGRP antagonist (gepant) 1 month prior to enrollment or during duration of study
* Use of verapamil during the study
* Use of CGRP monoclonal antibodies 3 months prior to enrollment or during duration of study.
* Subjects with a secondary cluster headache related to an underlying structural etiology identified by imaging (CT or MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in weekly frequency of cluster headache attacks | Baseline, week of treatment (days 1-7)
  Total number of cluster headache attacks experienced in one week

SECONDARY OUTCOMES:
Change in daily headache severity | Baseline, week of treatment (days 1-8)
  Change from baseline daily headache severity in days 1 through 8 in subjects treated with rimegepant, as measured on a Numeric Pain Rating Scale (NPRS), an 11-point scale from 0 to 10, where "0" indicates no pain and "10" suggests the most severe pain imaginable
Change in daily frequency of cluster headache attacks | Baseline, week of treatment (days 1-8)
  Total number of cluster headaches experienced daily

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Robertson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials